CLINICAL TRIAL: NCT02088307
Title: Evaluation of the Metabolic and Physiological Profiles of Patients Diagnosed With Cardiovascular Disease (CVD) Following Administration of the Novel Cardiovascular Vitamin, CardioLife
Brief Title: Study of the Cardiovascular Vitamin, CardioLife
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Anwar Tandar, Assistant Professor (Clinical), Division of Cardiology, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CARDIOLIFE--001
Record Dates: First submitted 2014-03-11; First posted 2014-03-14 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Cardiovascular Disease
Keywords: cardiovascular supplement; cardiovascular disease; coronary artery disease
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Subjects in the control arm will not receive an intervention.
- CardioLife (Experimental): The main ingredients in the CardioLife supplements are as follows: garlic, co-enzyme Q10, arjuna, hawthorn, guggul, red yeast rice, policosanol, nattokinase, tumeric/curcumin, ashwangandha, L-carnitine, grape seed extract and vitamin B12.
  Interventions: Dietary Supplement: CardioLife

INTERVENTIONS:
Dietary Supplement: CardioLife — Participants randomized to treatment arm will take dietary supplement as instructed.
  Arms: CardioLife

SUMMARY:
Evaluation of the metabolic and physiological characteristics of patients with diagnosed Cardiovascular Disease following administration of the Cardiovascular vitamin, CardioLife.

DETAILED DESCRIPTION:
The goal of this study is to evaluate the safety and efficacy of cardiovascular nutraceutical supplement, CardioLife™ in patients with diagnosed Cardiovascular Disease (CVD). CardioLife is a novel nutraceutical intended for the prevention and management of cardiovascular risk factors, enhancement of cardiac performance and the treatment of cardiac dysfunction. This is an oral vitamin supplement comprising of the following main ingredients: garlic co-enzyme Q10, Arjuna, Hawthorn, Guggul, Red Yeast Rice, Policosanol, Nattokinase, Tumeric/curcumin, ashangandha, L-carnitine, grape seed extract, and vitamin B12.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 90 years old and ability to understand the planned study.
* Patients with Cardiovascular Disease
* Able to comply with all study-related visits
* Able to give Informed Consent
* Negative for HcG with a serum pregnancy test
* If the patient has diabetes mellitus it must be controlled (HbA1c < 9.0%)
* Life expectancy of 1 year or more in the opinion of the investigator.
* Hematocrit ≥ 28.0%, White Blood Cell count ≤ 14,000, Platelet count ≥ 50,000, Serum bilirubin, ALT, AST x 2.5 time the upper level of normal.
* Controlled blood pressure (systolic blood pressure ≤160 and a diastolic blood pressure of ≤100 mmHG) and established anti-hypertensive therapy as necessary prior to entry into the study
* Patient must be on at least three of the listed medications for at least 30 days with no new medications to treat the disease introduced in the last month. Medications are: Anti-Platelet Therapy, Beta-Blockers, ACE/ARB, Calcium Blocker, Nitrates, After Load Reducing Agents, Lipid Lowering Agents, and/or Diuretics. Cardiac medications must be at stable doses with no dose change within the last 30 days.

Pre-existing condition (e.g. thromboembolic risk, diabetes, hypercholesterolemia are adequately controlled in the opinion of the investigator)

* Fertile patients (male and female) must agree to use an appropriate form of contraception while participating in the study.

Exclusion Criteria:

* Female who is pregnant or nursing, or of child bearing potential and is not using a reliable birth control method, or who intend to become pregnant during the tenure of this study.
* End stage renal disease (Creatinine ≤ 3.0 mg / dl) and/or dialysis
* Acute Myocardial Infarction 90 days prior to randomization.
* Inability or unwillingness to comply with the treatment protocol, follow-up, research tests, or give consent.
* Life expectancy <1 year due to concomitant illnesses
* Known cancer or malignancy within the last 5 years
* Prior admission for substance abuse
* Uncontrolled lipid levels as determined by the Investigator
* Untreated Hypothyroidism
* Known Congenital Heart Defects
* History of Ischemic and Non-Ischemic Cardiomyopathy or Heart Failure
* Body Mass Index (BMI) of 45 kg/m2 or greater
* Medication use of steroids 30 days prior to enrollment
* Current use of any Nutraceutical that contains ingredients known to affect blood pressure, or any active ingredients that are found in CardioLifeTM
* Patient receiving experimental medication or participating in another clinical study within 30 days of signing the informed consent
* In the opinion of the investigator or the sponsor, the patient is unsuitable for cellular therapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure | Baseline to 6 months

SECONDARY OUTCOMES:
Change in serum lipid levels | Baseline to 6 Months
Change plasma levels of endothelial progenitor cells (EPC) | Baseline to 6 Months
Change in cholesterol levels | 6 months
Change in homocysteine levels | 6 months
Change in erythrocyte sedimentation rate (ESR) levels | 6 months
Change in hs-C-reactive protein (CRP) levels | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Anwar Tandar, M.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah Hospitals and Clinics, Salt Lake City, Utah, United States